CLINICAL TRIAL: NCT06821581
Title: Economic-demographic Assessment of the Aseptic Mobilization of Knee Prostheses Through the RIPO Registry and Radiographic Analysis of the Case Series From the II Clinic of IOR
Acronym: AL-TKA
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Other Study IDs: AL-TKA
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Aseptic Loosening; Arthropathy of Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The increase in life expectancy is leading to an increase in the average age of patients undergoing total knee arthroplasty (TKA), and, consequently, an increase in the number of revisions. The main cause of TKA failure is aseptic mobilization, which is described as the loss of integration between the prosthetic component and the bone in the absence of infection. This represents a significant impact on professional and economic resources for the Italian healthcare system. Aseptic mobilization can be caused by inadequate initial fixation of the implant and/or mechanical or biological loss of fixation over time, factors that often occur simultaneously. A careful, methodical evaluation of post-operative radiographs of TKAs remains an important diagnostic tool. The analysis of the causes of aseptic mobilization of TKAs and the associated economic impact in the Emilia Romagna region is useful for providing an estimate of the problem and identifying potential areas for improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing knee prosthesis revision for aseptic mobilization
* Follow-up ≥ 2 years
* Willingness to participate in the study
* Both sexes
* Patients ≥ 18 years old

Exclusion Criteria:

* Patient refusal to participate in the study and sign the informed consent
* Simultaneous participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analysis will be conducted on implants performed in the Emilia-Romagna region from 2003 to 2022 and on implants performed at the II Orthopedic and Traumatological Clinic of the Rizzoli Orthopedic Institute during the same period
Sampling Method: Non-Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographic data | 24 months
  Collection of registry data related to the sample of patients undergoing TKA revision for aseptic mobilization, including demographic data

SECONDARY OUTCOMES:
Healthcare expenses | 24 months
  Collection of data related to healthcare expenses resulting from aseptic mobilization (TKA revision surgery, length of stay, 90-day readmission rate, any other hospitalizations, etc.)
Radiographic analysis | 24 months
  Radiographic analysis of the TKAs of patients who subsequently underwent revision surgery for aseptic mobilization at the II Orthopedic and Traumatological Clinic to assess the implant

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy